CLINICAL TRIAL: NCT05774236
Title: Cook´s Balloon Versus Dinoprostone for Labor Induction of Term Pregnancies With Fetal Growth Restriction (COLIGROW)
Brief Title: Cook´s Balloon Versus Dinoprostone for Labor Induction of Term Pregnancies With Fetal Growth Restriction
Acronym: COLIGROW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Ignacio Herraiz, Adjunct professor, Hospital Universitario 12 de Octubre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLIGROW; 2021-001726-22 (EudraCT Number); PI19_01005 (Other Grant/Funding Number: Instituto de Salud Carlos III); 2024-513523-16-00 (EU CTIS Number)
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Fetal Growth Retardation
Keywords: Fetal Growth Restriction; Cervical Ripening; Cook's Balloon; Dinoprostone; Labor Induction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Intervention Model Description: multicenter, randomized (1:1), open-label, 2-arm parallel group, controlled trial
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cook´s balloon (Experimental): Silicone 80 mL double-balloon cervical ripening catheter with an adjustable-length malleable stylet
  Interventions: Device: Cook´s balloon
- Vaginal dinoprostone (Active Comparator): Vaginal delivery system containing 10 mg dinoprostone (Prostaglandin E2) dispersed throughout its matrix and releasing approximately 0.3 mg/hour dinoprostone over a 24-hour period.
  Interventions: Drug: Vaginal dinoprostone

INTERVENTIONS:
Device: Cook´s balloon — Cervical ripening for induction of labor with a mechanical method (Cook´s balloon)
  Other Names: Cook® Cervical Ripening Balloon with Stylet; Double balloon catheter
  Arms: Cook´s balloon
Drug: Vaginal dinoprostone — Cervical ripening for induction of labor with a pharmacological method (vaginal dinoprostone)
  Other Names: Dinoprostone vaginal insert; Controlled-release dinoprostone delivery system; Vaginal prostaglandin E2
  Arms: Vaginal dinoprostone

SUMMARY:
The goal of this clinical trial is to compare how two methods for cervical ripening work in a population of singleton pregnancies with late-onset fetal growth restriction (FGR) at term.

The main question it aims to answer is whether Cook´s balloon (a mechanical method) is superior to vaginal dinoprostone (a pharmacological method) in achieving a vaginal delivery, without increasing neonatal morbidity.

Participants will be randomized to receive Cook´s balloon (experimental group) or vaginal dinoprostone (control group) for cervical ripening.

Researchers will compare both groups to see if Cook´s balloon is associated with a higher rate of vaginal delivery than vaginal dinoprostone and is not related to increased neonatal morbidity.

DETAILED DESCRIPTION:
Late-onset fetal growth restriction (FGR) represents the most common subtype of FGR (70-80%). The greatest risk for these fetuses appears once term pregnancy is reached, when stressful situations are added to their status of relative hypoxia, such as the appearance of contractions and funicular compression. Thus, it has been shown that from week 37-38 the risk of intrauterine mortality increases and there is a general consensus not to prolong these pregnancies beyond this period. In this situation, induction of labor is usually preferred over elective caesarean delivery. However, these fetuses have an increased risk of cesarean section for suspected fetal distress.

Mechanical methods for cervical ripening are associated with less uterine stimulation with a lower rate of tachysystole than prostaglandins. Therefore, these methods have been proposed as the optimal approach for late-onset FGR, since they could reduce the rate of cesarean sections for suspected fetal distress. However, there is no published randomized controlled trials on the use of different methods of cervical ripening for labor induction in late-onset FGR.

Thus, the investigators postulate that, in late-onset FGR, cervical ripening with a mechanical method (Cook´s balloon) achieves a higher percentage of vaginal deliveries than a pharmacological method (vaginal dinoprostone), being safe for both the mother and the newborn.

The main aim of this study is to evaluate whether cervical ripening with Cook balloon for labor induction at term gestation of singleton pregnancies with late-onset FGR achieves a higher rate of vaginal delivery compared to the use of vaginal dinoprostone, without increasing neonatal morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Age ≥ 18 years
* Gestational age (GA) dated by first trimester ultrasound ≥ 37+0 weeks
* Cephalic presentation
* Stage I fetal growth restriction, defined as the presence of at least one of these two criteria:

  1. Estimated fetal weight (EFW) < 3rd percentile
  2. EFW < 10th percentile and at least one of the following: 2.1) Umbilical artery pulsatility index > 95th percentile or 2.2) Cerebral-placental index < 5th percentile
* Bishop score < 7
* Intact fetal membranes
* No previous caesarean section
* No contraindications for vaginal delivery or labor induction.

Exclusion Criteria:

* Major fetal malformation
* Fetal genetic abnormality
* Fetal congenital infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Rate of vaginal delivery | 2 days (from admission to delivery)
  To assess whether cervical ripening with a Cook balloon for induction of labor of term pregnancies with FGR increases the rates of vaginal delivery with respect to the use of vaginal dinoprostone, without increasing neonatal morbidity.

SECONDARY OUTCOMES:
Rate of cesarean sections due to suspected fetal distress | 2 days (from admission to delivery)
  To assess whether cervical ripening with a Cook balloon for induction of labor of term pregnancies with FGR decreases the rates of cesarean sections due to suspected fetal distress with respect to the use of vaginal dinoprostone
Induction-to-delivery interval | 2 days (from admission to delivery)
  Comparison of the time interval between the onset of cervical ripening and delivery between the two arms
Neonatal morbidity | From delivery to discharge of the newborn (up to 1 month)
  To analyze the neonatal morbidity through the MAIN score (Morbidity assessment index for newborns) of neonatal morbidity and the duration of admissions to the Neonatal Intensive Care Unit (NICU).

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD that underlies the results reported in the publication will be shared after publications of primary results upon request of investigators whose proposed research has received IRB approval and after data use agreement
Supporting Information: Study Protocol
Time Frame: From the time of publication and for 5 years thereafter
Access Criteria: Upon request of investigators whose proposed research has received IRB approval and after data use agreement

REFERENCES:
- [Derived] Herraiz I, Meler E, Mazarico E, Bonacina E, Blanco JE, Villalain C, Barbero P, Peguero A, Barbera A, Sanchez ML, Llorente Munoz I, Lora Pablos D, Figueras F, Galindo A. Cook's balloon versus dinoprostone for Labour induction of term pregnancies with fetal GROWth restriction: study protocol for a randomised controlled trial in tertiary maternity hospitals in Spain (COLIGROW study). BMJ Open. 2024 Sep 30;14(9):e089628. doi: 10.1136/bmjopen-2024-089628. PMID 39349375